CLINICAL TRIAL: NCT04900870
Title: Evaluation of the Relationship Between Neck Pain and Temporomandibular Disorders in Office Workers
Status: Completed | Type: Observational
Sponsor: Tugba Sahbaz (Other)
Responsible Party: Sponsor-Investigator, Tugba Sahbaz, Director, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2021.03.114
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Neck Pain; Temporomandibular Disorder
Keywords: neck pain; temporomandibular disorder; office workers
MeSH Terms: conditions — Neck Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neck pain: Diagnostic Test: A self-administered questionnaire A self-administered questionnaire will be used to screen VAS scores, bournemouth neck questionnaire, demographic information and for temporomandibular pain Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments Axis I TMD Pain Screener, Symptom questionnaire and Axis II PHQ-4, Oral Behaviors Checklist .
- Neck pain with temeporomandibular pain: Diagnostic Test: A self-administered questionnaire A self-administered questionnaire will be used to screen VAS scores, bournemouth neck questionnaire, demographic information and for temporomandibular pain Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments Axis I TMD Pain Screener, Symptom questionnaire, Clinical Examination Form, Axis II Pain Drawing Graded Chronic Pain (version 2), JFLS-8 ,PHQ-4 Oral Behaviors Checklist.

SUMMARY:
The current study aimed to explore the associations between neck pain and temporomandibular disorders in office workers

DETAILED DESCRIPTION:
This is a cross-sectional study. All participants will provide informed consent before participating in the study. The study will be conducted in accordance with the Helsinki Declaration criteria. Data will be collected using questionnaires, which include information on demographic, clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55,
* Working on computer,
* Having neck pain at least three months.

Exclusion Criteria:

* Reporting pregnancy,
* Having a history of accidents,
* Trauma or surgery in the neck region and temporomandibular region,
* Congenital anomaly of the spine or temporomandibular joint,
* Rheumatologic disease,
* Osteoporosis,
* Spondylosis,
* Spondylolisthesis,
* Infection of the spine or temporomandibular joint
* Cervical disc herniation,
* Tumor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aged between 18 and 55, working on computer, having neck pain at least three months with or without temporomandibular pain
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Neck Bournemouth Questionnaire | 1 interview day
  The NBQ consists of 7 questions that examine the pain intensity, daily life activities, social activities, anxiety, emotional aspects of depression, kinesiophobia, and the ability to control pain. The items in the questionnaire are specific to patients with neck pain and each question evaluates a different parameter.The score for each measure are added. This can produce a value between a minimum score of 0, and a maximum score of 70. The higher the score reflects the degree of impact on a patient's life.
Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments | 1 interview day
  Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) is a dual-axis framework for the assessment and diagnosis of Axis I physical diagnoses for the most common TMDs and Axis II self-report psychosocial and behavioral screening questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Sahbaz, MD, Principal Investigator — University of Health Sciences, Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- University of Health Sciences, Kanuni Sultan Süleyman Training and Research Hospital,, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Selms MKA, Wiegers JW, van der Meer HA, Ahlberg J, Lobbezoo F, Visscher CM. Temporomandibular disorders, pain in the neck and shoulder area, and headache among musicians. J Oral Rehabil. 2020 Feb;47(2):132-142. doi: 10.1111/joor.12886. Epub 2019 Sep 24. PMID 31520546
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Kang JH. Effects on migraine, neck pain, and head and neck posture, of temporomandibular disorder treatment: Study of a retrospective cohort. Arch Oral Biol. 2020 Jun;114:104718. doi: 10.1016/j.archoralbio.2020.104718. Epub 2020 Apr 18. PMID 32334135
- [Background] Visscher CM, Schouten MJ, Ligthart L, van Houtem CM, de Jongh A, Boomsma DI. Shared Genetics of Temporomandibular Disorder Pain and Neck Pain: Results of a Twin Study. J Oral Facial Pain Headache. 2018 Spring;32(2):107-112. doi: 10.11607/ofph.2016. Epub 2018 Mar 6. PMID 29509827
- [Derived] Sahbaz T, Cigdem-Karacay B, Medin-Ceylan C, Korkmaz MD, Asik HK. The impact of self-reported temporomandibular pain on neck disability in office workers. J Back Musculoskelet Rehabil. 2025 Jul;38(4):774-782. doi: 10.1177/10538127251315829. Epub 2025 Mar 25. PMID 40129394